CLINICAL TRIAL: NCT03911856
Title: Unmasking Right Ventricular and Pulmonary Derangements With Exercise and Oxygen in Early Stage Cardiopulmonary Diseases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Bruce Johnson, Principal Investigator, Mayo Clinic
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 19-000626
Record Dates: First submitted 2019-04-05; First posted 2019-04-11 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Cardiopulmonary Disease
MeSH Terms: conditions — Pulmonary Heart Disease | interventions — Pulmonary Gas Exchange

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non-invasive assesment techniques (Experimental): We hypothesize that non-invasive indices of right ventricular RV (echocardiograph-derived strain and strain rate) and pulmonary (gas exchange-derived lung diffusion and surface area) function during light exercise will successfully identify and discern patients with known RV dysfunction pulmonary arterial hypertension and heart failure with preserved ejection fraction(PAH/HFpEF with RV failure) from those with known pulmonary dysfunction (PAH/HFpEF with pulmonary fibrosis). Additionally, we hypothesize that our assessment techniques will identify subtle derangements in RV and pulmonary function in newly diagnosed PAH and HFpEF patients, and that this may guide early and targeted therapeutic intervention.
  Interventions: Other: Echocardiography; Other: Pulmonary Gas Exchange
- Efficacy of acute-oxygen therapy during exercise (Experimental): We hypothesize that breathing hyperoxia will increase exercise capacity by reversing RV and pulmonary derangements, and that the mechanisms of action will be related to the underlying dysfunction (e.g., reducing pulse volume recording PVR, increasing RV functional reserve, increasing gas diffusion).
  Interventions: Other: Echocardiography; Other: Pulmonary Gas Exchange

INTERVENTIONS:
Other: Echocardiography — We hypothesize that non-invasive indices of RV (echocardiograph-derived strain and strain rate) and pulmonary (gas exchange-derived lung diffusion and surface area) function during light exercise will successfully identify and discern patients with known RV dysfunction (PAH/HFpEF with RV failure) from those with known pulmonary dysfunction (PAH/HFpEF with pulmonary fibrosis). Additionally, we hypothesize that our assessment techniques will identify subtle derangements in RV and pulmonary function in newly diagnosed PAH and HFpEF patients, and that this may guide early and targeted therapeutic intervention.
Other: Pulmonary Gas Exchange — We hypothesize that breathing hyperoxia will increase exercise capacity by reversing RV and pulmonary derangements, and that the mechanisms of action will be related to the underlying dysfunction (e.g., reducing PVR, increasing RV functional reserve, increasing gas diffusion).

SUMMARY:
Researchers are trying to develop innovative strategies that target the early identification heart and lung imbalances in patients with cardiopulmonary diseases.

ELIGIBILITY:
Inclusion criteria:

* Healthy controls (no known cardiac or pulmonary disease);
* PAH/HFpEF patients with known RV failure;
* PAH/HFpEF patients with known pulmonary failure
* Newly diagnosed PAH/HFpEF patients without any evidence of profound RV or pulmonary dysfunction.

Exclusion criteria:

* Persons unable to perform light exercise
* Persons pregnant or planning to be pregnant

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2020-01-09 (Actual); Primary Completion 2024-01-16 (Actual); Study Completion 2024-01-16 (Actual)

PRIMARY OUTCOMES:
Change in stroke volume (SV) during exercise and hyperoxia | 2 years
  Stroke volume will be measured with echocardiography at rest and during exercise while breathing room air and hyperoxia
Change in oxygen uptake (VO2) during exercise and hyperoxia | 2 years
  Oxygen uptake will be measured via pulmonary gas exchange at rest and during exercise while breathing room air and hyperoxia
Change in ventilatory efficiency (VE/VCO2) during exercise and hyperoxia | 2 years
  Ventilatory effciency will be measured via pulmonary gas exchange at rest and during exercise while breathing room air and hyperoxia

CONTACTS AND LOCATIONS:
Overall Officials: Bruce D Johnson, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials